CLINICAL TRIAL: NCT00006409
Title: Trial of Activity for Adolescent Girls (TAAG)
Acronym: TAAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, June Stevens, PhD, Distinguished Professor, Departments of Nutrition and Epidemiology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 934; U01HL066845 (NIH)
Record Dates: First submitted 2000-10-12; First posted 2000-10-13 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- School-based intervention (Experimental): TAAG health education included six lessons in each of 7th and 8th grades designed to enhance behavioral skills known to influence physical activity. TAAG physical education classes promoted moderate-vigorous physical activity for at least 50% of class time and encouraged teachers to promote physical activity outside of class. In conjunction with community partners, programs that were promoted outside of school included Dance Dance Revolution, after-school step aerobics class, before-school open gym, basketball camp, touch football, and weekend canoe programs. TAAG promotions used a social marketing approach to promote awareness of and participation in activities through media and promotional events.
  Interventions: Behavioral: Trial of Activity for Adolescent Girls (TAAG)
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Trial of Activity for Adolescent Girls (TAAG) — Intervention activities were designed to create (1) environmental and organizational changes supportive of physical activity and (2) cues, messages, and incentives to be more active. The intervention was designed to establish more opportunities, improve social support and norms, and increase self-efficacy, outcome expectations, and behavioral skills to foster greater moderate-vigorous physical activity (MVPA). An innovative feature of TAAG was linking school and community agencies to promote activity programs for girls. Finally, a TAAG Program Champion component was developed to foster sustainability after the 2-year staff-directed intervention. TAAG investigators recruited and trained Program Champions during the staff-directed intervention phase to promote maintenance of the program.
  Arms: School-based intervention

SUMMARY:
To test the effectiveness of a multicomponent school-based and community-linked intervention in preventing the decline in physical activity levels and cardiovascular fitness in girls in grades 6-8.

DETAILED DESCRIPTION:
BACKGROUND:

The Report of the Surgeon General on Physical Activity and Health (USDHHS, 1996) emphasized that regular physical activity has important health benefits including reducing the risk of heart disease, and helping to treat and prevent high blood pressure, high cholesterol, and diabetes, and to prevent osteoporosis and colon cancer. In addition, physical activity helps control weight, reduces feelings of depression and anxiety, and promotes psychological well being. Inactivity increases with age and is more common among women than men and among those with lower income, less education, and in minorities (USDHHS, 1996). Even though adolescents are more active than adults, many do not engage in recommended levels of physical activity, and participation declines with age throughout adolescence, especially in girls (USDHHS, 1996; CDC, 1997). Fourteen percent of teenage girls get no regular exercise, twice the percentage as for boys. The proportion of adolescent girls who participate in regular vigorous physical activity declines dramatically each year they are in high school, from 61 percent among 9th graders to 41percent among 12th grade girls. In high school, enrollment for girls in daily physical education classes dropped from 41 percent in 1991 to 25 percent in 1995. Both the CDC report (1997) and the Surgeon General's Report (USDHHS, 1996) recommended the need for research testing the effectiveness of a coordinated school-based physical activity intervention linked to community agency programs to increase physical activity by adolescent girls.

The study is the result of a Request for Applications released in January, 2000. Awards were made in September 2000.

DESIGN NARRATIVE:

The purpose of the multicenter randomized trial is to test the effectiveness of a multicomponent school-based and community-linked intervention in preventing the decline in physical activity levels and cardiovascular fitness in middle school girls (i.e., in grades 6-8). The interventions will provide skills-building, supportive environments, and opportunities for participation in physical activity during and outside of the school day. Phase 1 will be 24 months for protocol development and pilot work, Phase II is 44 months for two years of intervention and one year of follow-up, and Phase III is 4 months for close out of the Study Centers, and 16 months for the Coordinating Center to collaboratively analyze and report the results.

The randomized trial of 36 middle schools (6 per field site) will collect data by two-cross sectional samples, one taken at the sixth grade (at least 1,728 girls) in the Spring of 2003 and the other taken at the eighth grade (at least 3,456 girls) in the Spring of 2005. Follow-up data collection will also occur at the eighth grade in the Spring of 2006.

ELIGIBILITY:
School inclusion criteria:

* Public middle schools in which a majority of students lived in the surrounding community
* Enrollment of at least 90 8th-grade girls
* Yearly withdrawal rates less than 28%
* At least one semester of physical education required for each grade
* Willingness to sign a memorandum of understanding and accept random assignment of the school

Student exclusion criteria:

* Limited English-speaking skills
* Unable to participate in physical education classes due to a medical condition or disability
* Contraindications for participating in a submaximal exercise test

Ages: 12 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8727 (Actual)
Dates: Start 2000-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Elder, Principal Investigator — San Diego State University; Timothy Lohman, Principal Investigator — University of Arizona; Leslie Lytle, Principal Investigator — University of Minnesota; Russell Pate, Principal Investigator — University of South Carolina; June Stevens, Principal Investigator — University of North Carolina; Larry Webber, Principal Investigator — Tulane University; Deborah Young, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Murray DM, Catellier DJ, Hannan PJ, Treuth MS, Stevens J, Schmitz KH, Rice JC, Conway TL. School-level intraclass correlation for physical activity in adolescent girls. Med Sci Sports Exerc. 2004 May;36(5):876-82. doi: 10.1249/01.mss.0000126806.72453.1c. PMID 15126724
- [Background] Moody JS, Prochaska JJ, Sallis JF, McKenzie TL, Brown M, Conway TL. Viability of parks and recreation centers as sites for youth physical activity promotion. Health Promot Pract. 2004 Oct;5(4):438-43. doi: 10.1177/1524839903258222. PMID 15358916
- [Background] Stevens J, Murray DM, Catellier DJ, Hannan PJ, Lytle LA, Elder JP, Young DR, Simons-Morton DG, Webber LS. Design of the Trial of Activity in Adolescent Girls (TAAG). Contemp Clin Trials. 2005 Apr;26(2):223-33. doi: 10.1016/j.cct.2004.12.011. PMID 15837442
- [Background] Dishman RK, Motl RW, Sallis JF, Dunn AL, Birnbaum AS, Welk GJ, Bedimo-Rung AL, Voorhees CC, Jobe JB. Self-management strategies mediate self-efficacy and physical activity. Am J Prev Med. 2005 Jul;29(1):10-8. doi: 10.1016/j.amepre.2005.03.012. PMID 15958246
- [Background] Schmitz KH, Treuth M, Hannan P, McMurray R, Ring KB, Catellier D, Pate R. Predicting energy expenditure from accelerometry counts in adolescent girls. Med Sci Sports Exerc. 2005 Jan;37(1):155-61. doi: 10.1249/01.mss.0000150084.97823.f7. PMID 15632682
- [Background] Treuth MS, Schmitz K, Catellier DJ, McMurray RG, Murray DM, Almeida MJ, Going S, Norman JE, Pate R. Defining accelerometer thresholds for activity intensities in adolescent girls. Med Sci Sports Exerc. 2004 Jul;36(7):1259-66. PMID 15235335
- [Result] McMurray RG, Ring KB, Treuth MS, Welk GJ, Pate RR, Schmitz KH, Pickrel JL, Gonzalez V, Almedia MJ, Young DR, Sallis JF. Comparison of two approaches to structured physical activity surveys for adolescents. Med Sci Sports Exerc. 2004 Dec;36(12):2135-43. doi: 10.1249/01.mss.0000147628.78551.3b. PMID 15570151
- [Result] Birnbaum AS, Evenson KR, Motl RW, Dishman RK, Voorhees CC, Sallis JF, Elder JP, Dowda M. Scale development for perceived school climate for girls' physical activity. Am J Health Behav. 2005 May-Jun;29(3):250-7. doi: 10.5993/ajhb.29.3.6. PMID 15899688
- [Result] Catellier DJ, Hannan PJ, Murray DM, Addy CL, Conway TL, Yang S, Rice JC. Imputation of missing data when measuring physical activity by accelerometry. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S555-62. doi: 10.1249/01.mss.0000185651.59486.4e. PMID 16294118
- [Result] Voorhees CC, Murray D, Welk G, Birnbaum A, Ribisl KM, Johnson CC, Pfeiffer KA, Saksvig B, Jobe JB. The role of peer social network factors and physical activity in adolescent girls. Am J Health Behav. 2005 Mar-Apr;29(2):183-90. doi: 10.5993/ajhb.29.2.9. PMID 15698985
- [Result] Cohen DA, Ashwood S, Scott M, Overton A, Evenson KR, Voorhees CC, Bedimo-Rung A, McKenzie TL. Proximity to School and Physical Activity Among Middle School Girls: The Trial of Activity for Adolescent Girls Study. J Phys Act Health. 2006 Feb;3(s1):S129-S138. doi: 10.1123/jpah.3.s1.s129. PMID 28834509
- [Result] Cohen DA, Ashwood JS, Scott MM, Overton A, Evenson KR, Staten LK, Porter D, McKenzie TL, Catellier D. Public parks and physical activity among adolescent girls. Pediatrics. 2006 Nov;118(5):e1381-9. doi: 10.1542/peds.2006-1226. PMID 17079539
- [Result] Elder JP, Lytle L, Sallis JF, Young DR, Steckler A, Simons-Morton D, Stone E, Jobe JB, Stevens J, Lohman T, Webber L, Pate R, Saksvig BI, Ribisl K. A description of the social-ecological framework used in the trial of activity for adolescent girls (TAAG). Health Educ Res. 2007 Apr;22(2):155-65. doi: 10.1093/her/cyl059. Epub 2006 Jul 19. PMID 16855014
- [Result] Evenson KR, Birnbaum AS, Bedimo-Rung AL, Sallis JF, Voorhees CC, Ring K, Elder JP. Girls' perception of physical environmental factors and transportation: reliability and association with physical activity and active transport to school. Int J Behav Nutr Phys Act. 2006 Sep 14;3:28. doi: 10.1186/1479-5868-3-28. PMID 16972999
- [Result] Gittelsohn J, Steckler A, Johnson CC, Pratt C, Grieser M, Pickrel J, Stone EJ, Conway T, Coombs D, Staten LK. Formative research in school and community-based health programs and studies: "state of the art" and the TAAG approach. Health Educ Behav. 2006 Feb;33(1):25-39. doi: 10.1177/1090198105282412. PMID 16397157
- [Result] Grieser M, Vu MB, Bedimo-Rung AL, Neumark-Sztainer D, Moody J, Young DR, Moe SG. Physical activity attitudes, preferences, and practices in African American, Hispanic, and Caucasian girls. Health Educ Behav. 2006 Feb;33(1):40-51. doi: 10.1177/1090198105282416. PMID 16397158
- [Result] Lohman TG, Ring K, Schmitz KH, Treuth MS, Loftin M, Yang S, Sothern M, Going S. Associations of body size and composition with physical activity in adolescent girls. Med Sci Sports Exerc. 2006 Jun;38(6):1175-81. doi: 10.1249/01.mss.0000222846.27380.61. PMID 16775560
- [Result] McKenzie TL, Catellier DJ, Conway T, Lytle LA, Grieser M, Webber LA, Pratt CA, Elder JP. Girls' activity levels and lesson contexts in middle school PE: TAAG baseline. Med Sci Sports Exerc. 2006 Jul;38(7):1229-35. doi: 10.1249/01.mss.0000227307.34149.f3. PMID 16826019
- [Result] Moe SG, Pickrel J, McKenzie TL, Strikmiller PK, Coombs D, Murrie D. Using school-level interviews to develop a Multisite PE intervention program. Health Educ Behav. 2006 Feb;33(1):52-65. doi: 10.1177/1090198105282418. PMID 16397159
- [Result] Murray DM, Stevens J, Hannan PJ, Catellier DJ, Schmitz KH, Dowda M, Conway TL, Rice JC, Yang S. School-level intraclass correlation for physical activity in sixth grade girls. Med Sci Sports Exerc. 2006 May;38(5):926-36. doi: 10.1249/01.mss.0000218188.57274.91. PMID 16672847
- [Result] Saunders RP, Moody J. Community agency survey formative research results from the TAAG study. Health Educ Behav. 2006 Feb;33(1):12-24. doi: 10.1177/1090198105282410. PMID 16397156
- [Result] Staten LK, Birnbaum AS, Jobe JB, Elder JP. A typology of middle school girls: audience segmentation related to physical activity. Health Educ Behav. 2006 Feb;33(1):66-80. doi: 10.1177/1090198105282419. PMID 16397160
- [Result] Vu MB, Murrie D, Gonzalez V, Jobe JB. Listening to girls and boys talk about girls' physical activity behaviors. Health Educ Behav. 2006 Feb;33(1):81-96. doi: 10.1177/1090198105282443. PMID 16397161
- [Result] Young DR, Johnson CC, Steckler A, Gittelsohn J, Saunders RP, Saksvig BI, Ribisl KM, Lytle LA, McKenzie TL. Data to action: using formative research to develop intervention programs to increase physical activity in adolescent girls. Health Educ Behav. 2006 Feb;33(1):97-111. doi: 10.1177/1090198105282444. PMID 16397162
- [Result] Pfeiffer KA, Schmitz KH, McMurray RG, Treuth MS, Murray DM, Pate RR. Physical activities in adolescent girls: variability in energy expenditure. Am J Prev Med. 2006 Oct;31(4):328-31. doi: 10.1016/j.amepre.2006.06.002. Epub 2006 Aug 28. PMID 16979458
- [Result] Pate RR, Stevens J, Pratt C, Sallis JF, Schmitz KH, Webber LS, Welk G, Young DR. Objectively measured physical activity in sixth-grade girls. Arch Pediatr Adolesc Med. 2006 Dec;160(12):1262-8. doi: 10.1001/archpedi.160.12.1262. PMID 17146024
- [Result] Rushovich BR, Voorhees CC, Davis CE, Neumark-Sztainer D, Pfeiffer KA, Elder JP, Going S, Marino VG. The relationship between unsupervised time after school and physical activity in adolescent girls. Int J Behav Nutr Phys Act. 2006 Jul 31;3:20. doi: 10.1186/1479-5868-3-20. PMID 16879750
- [Result] Going S, Nichols J, Loftin M, Stewart D, Lohman T, Tuuri G, Ring K, Pickrel J, Blew R, J Stevens. Validation of bioelectrical impedance analysis (BIA) for estimation of body composition in Black, White and Hispanic adolescent girls. Int J Body Compos Res. 2006;4(4):161-167. PMID 17848976
- [Result] Nichols J, Going S, Loftin M, Stewart D, Nowicki E, Pickrel J. Comparison of two bioelectrical impedance analysis instruments for determining body composition in adolescent girls. Int J Body Compos Res. 2006;4(4):153-160. PMID 17607326
- [Result] Young DR, Felton GM, Grieser M, Elder JP, Johnson C, Lee JS, Kubik MY. Policies and opportunities for physical activity in middle school environments. J Sch Health. 2007 Jan;77(1):41-7. doi: 10.1111/j.1746-1561.2007.00161.x. PMID 17212759
- [Result] Saksvig BI, Catellier DJ, Pfeiffer K, Schmitz KH, Conway T, Going S, Ward D, Strikmiller P, Treuth MS. Travel by walking before and after school and physical activity among adolescent girls. Arch Pediatr Adolesc Med. 2007 Feb;161(2):153-8. doi: 10.1001/archpedi.161.2.153. PMID 17283300
- [Result] Evenson KR, Scott MM, Cohen DA, Voorhees CC. Girls' perception of neighborhood factors on physical activity, sedentary behavior, and BMI. Obesity (Silver Spring). 2007 Feb;15(2):430-45. doi: 10.1038/oby.2007.502. PMID 17299117
- [Result] Scott MM, Cohen DA, Evenson KR, Elder J, Catellier D, Ashwood JS, Overton A. Weekend schoolyard accessibility, physical activity, and obesity: the Trial of Activity in Adolescent Girls (TAAG) study. Prev Med. 2007 May;44(5):398-403. doi: 10.1016/j.ypmed.2006.12.010. Epub 2006 Dec 29. PMID 17292958
- [Result] Loftin M, Nichols J, Going S, Sothern M, Schmitz KH, Ring K, Tuuri G, Stevens J. Comparison of the validity of anthropometric and bioelectric impedance equations to assess body composition in adolescent girls. Int J Body Compos Res. 2007;5(1):1-8. PMID 18163160
- [Result] Scott MM, Evenson KR, Cohen DA, Cox CE. Comparing perceived and objectively measured access to recreational facilities as predictors of physical activity in adolescent girls. J Urban Health. 2007 May;84(3):346-59. doi: 10.1007/s11524-007-9179-1. PMID 17401691
- [Result] Treuth MS, Catellier DJ, Schmitz KH, Pate RR, Elder JP, McMurray RG, Blew RM, Yang S, Webber L. Weekend and weekday patterns of physical activity in overweight and normal-weight adolescent girls. Obesity (Silver Spring). 2007 Jul;15(7):1782-8. doi: 10.1038/oby.2007.212. PMID 17636097
- [Result] Dowda M, McKenzie TL, Cohen DA, Scott MM, Evenson KR, Bedimo-Rung AL, Voorhees CC, Almeida MJ. Commercial venues as supports for physical activity in adolescent girls. Prev Med. 2007 Aug-Sep;45(2-3):163-8. doi: 10.1016/j.ypmed.2007.06.001. Epub 2007 Jun 7. PMID 17673281
- [Derived] Budd EL, McQueen A, Eyler AA, Haire-Joshu D, Auslander WF, Brownson RC. The role of physical activity enjoyment in the pathways from the social and physical environments to physical activity of early adolescent girls. Prev Med. 2018 Jun;111:6-13. doi: 10.1016/j.ypmed.2018.02.015. Epub 2018 Feb 12. PMID 29447926
- [Derived] Webber LS, Catellier DJ, Lytle LA, Murray DM, Pratt CA, Young DR, Elder JP, Lohman TG, Stevens J, Jobe JB, Pate RR; TAAG Collaborative Research Group. Promoting physical activity in middle school girls: Trial of Activity for Adolescent Girls. Am J Prev Med. 2008 Mar;34(3):173-84. doi: 10.1016/j.amepre.2007.11.018. PMID 18312804

RESULTS

PARTICIPANT FLOW:
Groups:
- 6th-grade/2003 - Intervention: Cross-sectional sample of 6th-grade girls in schools that were randomized to receive the intervention (data collected at baseline)
- 6th-grade/2003 - Control: Cross-sectional sample of 6th-grade girls in schools that were randomized to not receive the intervention (data collected at baseline)
- 8th-grade/2005 - Intervention: Cross-sectional sample of 8th-grade girls in schools that were randomized to receive the intervention (data collected after 2 years of intervention, including "baseline" data reported here)
- 8th-grade/2005 - Control: Cross-sectional sample of 8th-grade girls in schools that were randomized to not receive the intervention (data collected after 2 years of intervention, including "baseline" data reported here)
- 8th-grade/2006 - Intervention: Cross-sectional sample of 8th-grade girls in schools that were randomized to receive the intervention (data collected after 3 years of intervention, including "baseline" data reported here)
- 8th-grade/2006 - Control: Cross-sectional sample of 8th-grade girls in schools that were randomized to not receive the intervention (data collected after 3 years of intervention, including "baseline" data reported here)
Period: Baseline
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control
Started | 865 | 856 | 0 | 0 | 0 | 0
Completed | 817 | 786 | 0 | 0 | 0 | 0
Not Completed | 48 | 70 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 48 | 70 | 0 | 0 | 0 | 0
Period: Post-2 Year Intervention
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control
Started | 0 (6th grade/2003 sample was not followed over time) | 0 (6th grade/2003 sample was not followed over time) | 1791 (Sample is independent of 6th-grade/2003 sample that was measured at baseline) | 1713 (Sample is independent of 6th-grade/2003 sample that was measured at baseline) | 0 | 0
Completed | 0 | 0 | 1540 | 1545 | 0 | 0
Not Completed | 0 | 0 | 251 | 168 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 251 | 168 | 0 | 0
Period: Post-3 Year Intervention
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control
Started | 0 | 0 | 0 (8th-grade/2005 sample was not followed over time) | 0 (8th-grade/2005 sample was not followed over time) | 1726 (Sample is independent of 8th-grade/2005 sample that was measured post-2 year intervention) | 1776 (Sample is independent of 8th-grade/2005 sample that was measured post-2 year intervention)
Completed | 0 | 0 | 0 | 0 | 1664 | 1714
Not Completed | 0 | 0 | 0 | 0 | 62 | 62
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 62 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control | Total
Number analyzed (Participants) | 865 | 856 | 1791 | 1713 | 1726 | 1776 | 8727
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 865 | 856 | 1791 | 1713 | 1726 | 1776 | 8727
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.94 (0.49) | 11.98 (0.55) | 14.00 (0.53) | 13.99 (0.52) | 13.97 (0.49) | 13.99 (0.49) | 11.96 (0.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 865 | 856 | 1791 | 1713 | 1726 | 1776 | 8727
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: MET-weighted MVPA: Daily Minutes of Moderate-to-vigorous Physical Activity (MVPA) Weighted by Metabolic Equivalent of Task (MET)
Time Frame: Post-2 year intervention
Measure: Mean (Standard Error); unit: Minutes of MET-weighted MVPA˙
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control
Number analyzed (Participants) | 0 | 0 | 1540 | 1545 | 0 | 0
Minutes of MET-weighted MVPA˙ |  |  | 136.5 (5.16) | 136.9 (5.16) |  |

2. Primary Outcome: MET-weighted MVPA: Daily Minutes of Moderate-to-vigorous Physical Activity (MVPA) Weighted by Metabolic Equivalent of Task (MET)
Time Frame: Post-3 year intervention
Measure: Mean (Standard Error); unit: Minutes of MET-weighted MVPA˙
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1664 | 1714
Minutes of MET-weighted MVPA˙ |  |  |  |  | 136.4 (7.31) | 125.5 (7.31)

ADVERSE EVENTS:
Arm/Group | 6th-grade/2003 - Intervention | 6th-grade/2003 - Control | 8th-grade/2005 - Intervention | 8th-grade/2005 - Control | 8th-grade/2006 - Intervention | 8th-grade/2006 - Control
Serious Adverse Events (participants affected / at risk) | 0/865 | 0/856 | 0/1791 | 0/1713 | 0/1726 | 0/1776
Other Adverse Events (participants affected / at risk) | 0/865 | 0/856 | 0/1791 | 0/1713 | 0/1726 | 0/1776

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No